CLINICAL TRIAL: NCT00671216
Title: A Single Centre, Randomised, Placebo-controlled, Four-way Cross Over Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK233705 and GW642444 as Monotherapies and in Combination in Healthy Subjects.
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Inhaled Doses of GSK233705 and GW642444 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DB1111509
Record Dates: First submitted 2008-04-30; First posted 2008-05-05 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: safety; pharmacodynamics; Muscarinic Receptor Antagonist; tolerability; healthy subjects; GS642444; GSK233705; Anticholinergic; ß2 agonist; pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Period 1 (Experimental): Subjects will receive first placebo, then GSK233705, GW642444 and combination of GSK233705 and GW642444
  Interventions: Drug: GSK233705; Drug: GW642444; Drug: GSK233705 and GW642444; Drug: Placebo
- Period 2 (Experimental): Subjects will receive first combination of GSK233705 and GW642444, then placebo, GSK233705 and GW642444
  Interventions: Drug: GSK233705; Drug: GW642444; Drug: GSK233705 and GW642444; Drug: Placebo
- Period 3 (Experimental): Subjects will receive first GSK233705, then GW642444, combination of GSK233705 and GW642444 and later placebo
  Interventions: Drug: GSK233705; Drug: GW642444; Drug: GSK233705 and GW642444; Drug: Placebo
- Period 4 (Experimental): Subjects will receive first GW642444, then combination of GSK233705 and GW642444, placebo, and later GSK233705
  Interventions: Drug: GSK233705; Drug: GW642444; Drug: GSK233705 and GW642444; Drug: Placebo

INTERVENTIONS:
Drug: GSK233705 — Subjects will receive 200 (mcg) microgram once daily as a single dose
Drug: GW642444 — Subjects will receive 50 mcg once daily as a single dose
  Other Names: GSK233705
Drug: GSK233705 and GW642444 — Subjects will receive combination of GSK233705 200 mcg and GW642444 50 mcg as a single oral dose
Drug: Placebo — Placebo matching study medication will be inhaled by subjects

SUMMARY:
GW642444 and GSK233705 are in development for treatment of Chronic Obstructive Pulmonary Disease. Development of these two inhaled drugs as a combination therapy would have potential for improved patient benefit as they both work through different mechanisms and the combined bronchodilatory effect might be additive. This study will look at the this combination, for the first time, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 65 years of age.
* Female subjects must be of non childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal
* Male subjects must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until 90 days post-last dose.
* BMI within the range 18 - 30 kg/m2 (inclusive).
* Average QTc(B)≤450 msec taken from triplicate assessments at screening.
* No clinically active and relevant abnormality on 12-lead ECG at screening or 24h Holter ECG.
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Available to complete the study

Exclusion Criteria:

* Any clinically important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead). 24hr Holter monitoring outside normal limits.
* A history of breathing problems (i.e. history of asthmatic symptomatology, unless asthma in childhood that has now resolved and no longer requires maintenance therapy which should not be an exclusion).
* A mean QTc(B) value at screening >450msec, or an ECG that is not suitable for QT measurements (e.g. LBBB or poorly defined termination of the T wave).
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening.
* A mean heart rate outside the range 40-90 bpm at screening.
* The subject has a positive pre-study drug/alcohol screen. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody (if determined by the local SOP's).
* History of high alcohol consumption within 3months of the study defined as:
* an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, (except for simple analgesics eg paracetamol), including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products prior to screening.
* The subject is unable to use the novel dry powder inhaler correctly.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, Tiotropium, atropine and any of its derivatives.
* Any adverse reaction including immediate or delayed hypersensitivity to any β2 agonist or sympathomimetic drug,
* The subject has a known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and MgSt.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-05-20 (Actual); Primary Completion 2008-07-07 (Actual); Study Completion 2008-07-07 (Actual)

PRIMARY OUTCOMES:
General safety endpoints: measured over 24 hours post dose for all 4 dose periods, heart rate, systolic and diastolic blood pressure, 12- lead ECG and lung function and clinical laboratory safety tests. Adverse events over whole study. | Up to Day 2

SECONDARY OUTCOMES:
Blood levels of GW642444, Blood levels of GSK233705, Blood Levels of potassium | Pre-dose; Day 1- 5, 15 and 30 minutes, 1, 2, 4, 5,6, 8, 12, 16 and 24 hours and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing the attached study results summary.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study DB1111509 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/DB1111509?search=study&search_terms=DB1111509#rs
- Available data/document: Individual Participant Data Set: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: DB1111509 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register